CLINICAL TRIAL: NCT05494762
Title: A Phase 1a/1b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-B167, Alone and in Combination With Tislelizumab in Patients With Selected Advanced or Metastatic Solid Tumors
Brief Title: Safety, Pharmacokinetics, and Antitumor Activity of BGB-B167 Alone and in Combination With Tislelizumab (BGB-A317) in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-B167-101
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): Part A: Increasing dose levels of BGB-B167 monotherapy; Part B: Increasing dose levels of BGB-B167 in combination with tislelizumab (BGB-A317)
  Interventions: Drug: BGB-B167; Drug: Tislelizumab
- Phase 1b: Dose Expansion (Experimental): BGB-B167 alone or in combination with tislelizumab (BGB-A317)
  Interventions: Drug: BGB-B167; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-B167 — Intravenous administration
Drug: Tislelizumab — Intravenous administration
  Other Names: BGB-A317

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of BGB-B167 monotherapy and in combination with tislelizumab (BGB-A317) in participants with select advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Participants with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors previously treated with standard systemic therapy or for whom treatment is not available, not tolerated, or refused, or not expected to provide significant clinical benefit or be tolerated in the medical judgement of the investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Adequate organ function as indicated by laboratory values during screening or ≤ 7 days before the first dose of study drug(s)

Exclusion Criteria:

* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent
* History of severe hypersensitivity reactions to other monoclonal antibody products or their excipients
* Women who are pregnant or are breastfeeding

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 3 years
Phase 1a: Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to approximately 3 years
Phase 1a: Number of Participants Experiencing AEs Meeting Protocol-defined Dose-limiting Toxicity (DLT) Criteria | Up to approximately 3 years
Phase 1a: Maximum tolerated dose (MTD) | Up to approximately 3 years
  MTD is defined as the highest tolerated dose with the target toxicity rate of 30%
Phase 1a: Recommended Phase 2 doses (RP2Ds) | Up to 90 days after the last dose of study drug(s); up to approximately 3 years
  RP2Ds of BGB-B167 alone or in combination with tislelizumab will be determined based on a biologically effective dose
Phase 1b: Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as determined by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to approximately 3 years
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as determined by investigators per RECIST v1.1
Phase 1a and 1b: Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from the first determination of a confirmed objective response until the first documentation of progression or death due to any cause, whichever occurs first, as determined by investigators per RECIST v1.1
Phase 1a and 1b: Disease Control Rate (DCR) | Up to approximately 3 years
  DCR is defined as the percentage of participants with best overall response (BOR) of confirmed CR, PR, or stable disease, as determined by investigators per RECIST v1.1
Phase 1a and 1b: Clinical Benefit Rate (CBR) | Up to approximately 3 years
  CBR is defined as the percentage of patients with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks, as determined by investigators per RECIST v1.1
Phase 1b: Progression-free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from the date of the first administration of study drug to the date of the first documentation of disease progression or death due to any cause, whichever occurs first, as determined by investigators per RECIST v1.1
Phase 1a and 1b: Serum Concentration of Tislelizumab | Up to approximately 3 years
Phase 1a and 1b: Maximum observed serum concentration (Cmax) of BGB-B167 | Up to approximately 3 years
Phase 1a and 1b: Minimum observed serum concentration (Cmin) of BGB-B167 | Up to approximately 3 years
Phase 1a and 1b: Time to reach maximum observed serum concentration (Tmax) of BGB-B167 | Up to approximately 3 years
Phase 1a and 1b: Elimination half life (t1/2) of BGB-B167 | Up to approximately 3 years
Phase 1a and 1b: Area under the concentration-time curve in 1 dosing interval (AUCtau) of BGB-B167 | Up to approximately 3 years
Phase 1a and 1b: Total body clearance (CL) of BGB-B167 | Up to approximately 3 years
Phase 1a and 1b: Volume of distribution at steady state (Vss) of BGB-B167 | Up to approximately 3 years
Phase 1b: Number of Participants with AEs or SAEs | Up to approximately 3 years
Phase 1a and 1b: Number of Participants with Antidrug Antibodies (ADAs) | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (8):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
- Australia (5):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/